CLINICAL TRIAL: NCT01953237
Title: MedActive: A Smartphone Intervention to Improve Adherence to Antipsychotic Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Julie Kreyenbuhl, Associate Professor of Psychiatry, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HP-00059272
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; antipsychotic medication adherence; mobile phones
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Individuals randomized to the control condition will be provided with a smartphone free of charge with unlimited use of the phone's voice and internet capabilities. All participants randomized to this condition will also have their antipsychotic medication adherence assessed over the 3-month period. All participants will be contacted by research staff to trouble-shoot problems with the smartphone at the end of the first week, but will receive no additional contact from research staff until the end of the trial.
  Interventions: Device: Smartphone
- MedActive (Experimental): Participants randomized to the MedActive condition will complete a 1-hour training session on MedActive, which will include ascertaining their antipsychotic administration schedule that will be pre-programmed into the application along with other personalized features. Each participate will be asked to use the medActive application over the following three months. All participants randomized to this condition will also have their antipsychotic medication adherence assessed over the 3-month period.
  Interventions: Behavioral: MedActive

INTERVENTIONS:
Behavioral: MedActive — Participants randomized to the MedActive condition will complete a 1-hour training session on MedActive, which will include ascertaining their antipsychotic administration schedule that will be pre-programmed into the application along with other personalized features. Each participate will be asked to use the medActive application over the following three months. All participants randomized to this condition will also have their antipsychotic medication adherence assessed over the 3-month period.
  Arms: MedActive
Device: Smartphone
  Arms: Control

SUMMARY:
We propose to develop and pilot test the effect of a mobile smartphone intervention, MedActive, on improving antipsychotic adherence among individuals with schizophrenia.

DETAILED DESCRIPTION:
Up to 60% of individuals with schizophrenia do not take their antipsychotic medications as prescribed, which can lead to symptom relapse, decreased functioning, hospitalization, and increased healthcare costs. Recent studies of both patient- and pharmacy-based interventions utilizing behavioral tailoring, environmental supports, and medication monitoring have shown promise in improving antipsychotic adherence. However, there is continued need for effective adherence-enhancing interventions (AEIs) that are less resource intensive and more widely accessible by the broad range of individuals in need of assistance with medication management. Over the last decade, technological advances in internet and cellular communication, including the emergence of mobile 'smartphones', have revolutionized the way our society communicates. Whereas a variety of mobile phone-based applications have been shown to be effective for improving health outcomes such as medication adherence for a number of medical conditions, few such applications have been developed for individuals with schizophrenia. Therefore, in response to NIMH PAR-09-173, we propose to develop and pilot test the effect of a mobile smartphone intervention, MedActive, on improving antipsychotic adherence among this population. We used the Information-Motivation-Behavioral (IMB) Skills Model of adherence as the theoretical framework to inform the conceptualization of MedActive. The IMB Skills Model posits that individuals who are well-informed and motivated to adhere will enact adherence-related behavioral skills that lead to adherence behaviors and favorable health outcomes. MedActive will provide personalized reminders to patients to take their antipsychotic medications as prescribed and will query them about their intentions to take the medication, the occurrence of side effects, and the presence of positive psychotic symptoms. Summaries of these ecological momentary assessments of adherence, symptoms, and side effects will be made available to the individual on the phone and to their psychiatrist through a secure, online clinician interface. Using an iterative user-centered design approach, the specific aims of this proposal are to (1) collaborate with individuals with schizophrenia, psychiatrists and an expert advisory group to develop the initial version of MedActive; (2) conduct laboratory usability testing and a short-term field trial in 10 individuals with schizophrenia and their psychiatrists to determine the preliminary acceptability and feasibility of MedActive in clinical practice; and (3) conduct a randomized pilot trial of MedActive compared to providing a smartphone alone in 40 individuals with schizophrenia and their psychiatrists to evaluate its effect on antipsychotic adherence. We will also explore whether psychiatric symptoms and neuropsychological impairments moderate the effect of MedActive on adherence. If shown to be effective, MedActive will introduce a paradigm shift in medication self-management by individuals with schizophrenia and in treatment monitoring by their clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Decisional capacity to provide informed consent
* Chart diagnosis of schizophrenia or schizoaffective disorder
* Currently prescribed at least one oral antipsychotic medication
* Self administers at least one oral antipsychotic medication
* 18-64 years of age
* English Speaking
* Be able to read English

Exclusion Criteria:

* Has visual, hearing, voice, or motor impairment that would prevent completion of study procedures or use of mobile phone

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Kreyenbuhl, Pharm.D PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- Outpatient clinics within the University of Maryland Division of Community Psychiatry, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | MedActive
Started | 10 | 21
Completed | 10 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | MedActive | Total
Number analyzed (Participants) | 10 | 21 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (12.9) | 49.5 (10.2) | 48.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 6 | 12 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 0 | 2 | 2
  Race: Black or African American | 10 | 18 | 28
  Race: Multiple races | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Antipsychotic Medications
Description: A measure of the extent to which participants self-reported taking their antipsychotic medications as prescribed
Time Frame: 3 month period
Measure: Mean (Standard Deviation); unit: percentage of days adherent
Arm/Group | Control | MedActive
Number analyzed (Participants) | 10 | 21
percentage of days adherent | 92.6 (10.6) | 93.4 (10.3)
Statistical Analysis 1: Comparison: Control vs MedActive; Test type: Superiority or Other; p = 0.5580, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Control | MedActive
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/21
Other Adverse Events (participants affected / at risk) | 0/10 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No